CLINICAL TRIAL: NCT02929368
Title: Randomized Controlled Noninferiority Study to Evaluate Safety and Efficacy of the Integrated Magnetic Tracking and ECG-guided Tip Location System (SHERLOCK 3CG) vs. Fluoroscopy in Implantation of Peripherally Inserted Central Catheter
Brief Title: SHERLOCK 3CG vs. Fluoroscopy in Implantation of PICC-Line
Acronym: 3CG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jena University Hospital (Other)
Responsible Party: Principal Investigator, Ulf Teichgräber, Director of Radiology Department, Jena University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4567/10/15
Record Dates: First submitted 2016-07-01; First posted 2016-10-11 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Patients With PICC-Line
Keywords: PICC-Line

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluoroscopy (Active Comparator): PICC Implantation under x-ray
  Interventions: Device: PICC implantation under fluoroscopy
- Sherlock System (BARD) (Active Comparator): PICC Implantation with Integrated Magnetic Tracking and ECG-guided Tip Location System
  Interventions: Device: PICC Implantation under Sherlock System

INTERVENTIONS:
Device: PICC implantation under fluoroscopy — PICC Catheter implantation
  Arms: Fluoroscopy
Device: PICC Implantation under Sherlock System — PICC Catheter implantation
  Arms: Sherlock System (BARD)

SUMMARY:
Peripherally inserted central catheters, or PICC lines, has now been successfully in use for many years, especially in the chemotherapeutic treatment of oncologic patients or in parenertal nutrition. The implantation of PICC lines is mostly performed under x-ray (fluoroscopy). The aim of the clinical study is to assess the safety and the efficacy of the SHERLOCK-Systems eliminating the confirmatory chest x-ray exposure. Additionally, the SHERLOCK-System immediately confirms the PICC tip position even at the bedside of the patient, thus, saving costs and time.

DETAILED DESCRIPTION:
Peripherally inserted central catheters, or PICC lines, are clinically used for many years in the treatment of patients, whereby the implantation occurs under x-ray/fluoroscopy. Female and male patients of legal age that have the medical indication for Power-PICC-Line catheter implantation can be screened for the study. These medical indications include the necessity of chemotherapy in the course of an oncological treatment or parenteral nutrition. The study objective is to test the efficacy and safety of the SHERLOCK system, evaluated by a monocentric, randomized-controlled study. The advantage for the participating patients lies in a reduced radiation exposure due to the discontinued final chest x-ray examination (fluoroscopy). Furthermore, the SHERLOCK system can be deployed directly on ward, at the patient's bedside leading to a cost and time saving. Recruited in- and outpatients (of legal age) with indication for Power-PICC-Line catheter implantation will be randomly assigned to one of the two arms (fluoroscopy or SHERLOCK). Depending on randomization, the Power-PICC implantation occurs either under fluoroscopy or with the SHERLOCK system. All related substances, measures or procedures are performed according to the clinical routine. The medical device is a fully integrated magnetic tracking and ECG-based peripherally inserted central catheter (PICC) tip confirmation technology applied on patients with normal sinus rhythm and placed through a peripheral vein. The Sherlock system is CE-certified since December 2011.

The referral of patients with indication to PICC-Line implantation at the institute of diagnostic and interventional radiology occurs through different departments of the University Hospital Jena. The patients are registered for radiological treatment and checked again by a radiologist if a PICC-Line implantation is indicated. If this is the case, the radiologist conducts an informed consent discussion with the patient about possible complications and risks during intervention and informs him also about a possible study. After signature of the written informed consent, the patient is included. On the intervention day, the patient is randomly assigned to one of the two study arms through RandomTool (Sherlock vs. fluoroscopy). According to randomization group, the PICC catheter is implanted (duration: 30 minutes) and eventually a chest x-ray (fluoroscopy) is performed to assess safety and efficacy.The intervention time from puncture to catheter placement is documented. After intervention, the patient is transferred back to the ward or sent home in hemodynamically stable conditions. The examination of the puncture site before discharge is performed by a ward physician or by the family doctor. 24 h after PICC-Line implantation, the treating physician is contacted and questioned about possible complications (catheter occlusion, haematoma, infection of the puncture site, arm vein thrombosis, pain, etc.), that are then thoroughly documented.

ELIGIBILITY:
Inclusion Criteria:

* female, male
* adults ≥ 18 years
* medical indication for Power-PICC-Line catheter implantation because of chemotherapy or parenertal nutrition
* in- and outpatients

Exclusion Criteria:

* children and adolescents < 18 years
* systemic or local infection of the interventional location
* known allergy to used material
* general contraindication of Power-PICC-Line catheter implantation
* nonexistent sinus rhythm (5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2016-06; Primary Completion 2018-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Tip Placement efficiency measured by chest radiograph | through study completion, an average of 2 years
  Corect placement through anatomic evaluation of chest x-ray measuring catheter tip max. two vertebral bodies under carina

SECONDARY OUTCOMES:
Safety measured by follow-up interview with referring physician and documentation of AE | Follow-up within one week
  Documentation of periprocedural complications
Implantation time | intraoperative
  time during PICC implantation

CONTACTS AND LOCATIONS:
Overall Officials: Heike Habrecht, Dr. med., Principal Investigator — University Hospital Jena, Germany
Locations (1):
- University Hospital Jena, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mack V, Nissler D, Kasikci D, Malouhi A, Aschenbach R, Teichgraber U. Magnetic Tracking and Electrocardiography-Guided Tip Confirmation System Versus Fluoroscopy for Placement of Peripherally Inserted Central Catheters: A Randomized, Noninferiority Comparison. Cardiovasc Intervent Radiol. 2020 Dec;43(12):1891-1897. doi: 10.1007/s00270-020-02551-0. Epub 2020 Jun 17. PMID 32556606